CLINICAL TRIAL: NCT03529448
Title: Phase Ib, Open-label, Multicenter, Intrapatient Dose-escalation Clinical Trial to Assess the Safety Profile of the TN-TC11G (THC+CBD) Combination With Temozolomide and Radiotherapy in Patients With Newly-diagnosed Glioblastoma
Brief Title: TN-TC11G (THC+CBD) Combination With Temozolomide and Radiotherapy in Patients With Newly-diagnosed Glioblastoma
Acronym: GEINOCANN
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Grupo Español de Investigación en Neurooncología (Other)
Collaborators: Medical Cannabis Bike Tour (Unknown); Voices Against Brain Cancer (Unknown); Tilray (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GEINO-1601; 2016-003216-12 (EudraCT Number)
Record Dates: First submitted 2018-04-23; First posted 2018-05-18 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Glioblastoma
Keywords: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Phase Ib, intra-patient dose escalation trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TN-TC11G, radiotherapy and Temozolomide Oral Product (Experimental): During Phase Ib, Four to seven weeks after surgical diagnosis, concurrent with radiotherapy (STUPP)
  + temozolomide (75mg/m2/day for 42 days) +TN-TC11G will be evaluated. During radiation therapy, temozolomide and TN-TC11G will be administered. This last, as the dose that have been selected previously, based on dose-titration period. Patient specific dose will remain until progresion of disease, unacceptable toxicity, non-compliance, consent withdrawal up to 2 years.
  Interventions: Drug: TN-TC11G; Drug: Temozolomide Oral Product; Radiation: Radiotherapy

INTERVENTIONS:
Drug: TN-TC11G — TN-TC11G dose will be gradually increased as follows:
  Week 1: TN-TC11G: 0-0-5 mg (THC 5 mg + CBD 5 mg; in the mornings, 90 minutes after breakfast; in the afternoons, 90 minutes after lunch; in the evenings, 90 minutes after dinner).
  Week 2: TN-TC11G: 5-0-5 mg Week 3: TN-TC11G: 5-5-5 mg Week 4: TN-TC11G: 5-5-10 mg Week 5: TN-TC11G: 5-5-15 mg Week 6: TN-TC11G: 10-10-15 mg Week 7: TN-TC11G: 10-10-20 mg. Week 8: TN-TC11G: 15-15-30 mg Week 9: TN-TC11G: 20-20-40 mg TN-TC11G will be administered daily at the relevant dose level according to the individual titration performed in the first 9 weeks of treatment. If there is any dose reduction, the reduced dose must be administered.
Drug: Temozolomide Oral Product — During RT, patients will receive Temozolomide (TMZ). All patients will be given TMZ at 75 mg/m2/d concurrently with RT for a maximum of 42 days.
  At 4 weeks after RT completion, patients will start taking TMZ at 150 mg/m2/d for the first 5 days of a 28-day cycle. If first cycle is well tolerated, patients will receive TMZ at 200 mg/m2/d for the first 5 days of every subsequent 28-day cycle for another 5 cycles.
  Other Names: Temozolomide
Radiation: Radiotherapy — All the patients will receive the Stupp regimen. The radiotherapy (RT) treatment will be administered in fractions of 1.8-2.0 Gy/day delivered 5 days/week to a total dose of 58-60 Gy. Radiotherapy will be delivered to the gross tumor volume with a 2-3 cm margin for the clinical target volume.
  Other Names: STUPP

SUMMARY:
Glioblastoma is the primary brain tumour with the worst prognosis: median survival is only 12 months despite the use of the most advanced treatments. In the past 10 years, survival in the treatment of this disease has not advanced significantly, with the postoperative standard being the administration of chemoradiotherapy with temozolomide, followed by 6 cycles of sequential chemotherapy with temozolomide.

Δ9-tetrahydrocannabinol (THC) and cannabidiol (CBD) have shown a clear synergistic antitumour effect with temozolomide and radiotherapy in preclinical glioma models. THC and CBD have a wide variety of biological effects by binding with and activating the type 1 and type 2 cannabinoid receptors (CB1 expressed in certain neuronal areas of the brain and CB2 expressed in the immune system and in glial cells). The activation of these receptors initiates a signalling pathway, called the endoplasmic reticulum stress response, which generates tumour cell autophagy by activating TRB3.

Given these data, the Spanish Group for Neuro-oncology (GEINO) proposes developing a phase Ib, open-label, multicenter, intrapatient dose-escalation clinical trial to assess the safety profile of the THC+CBD combination at a 1:1 ratio, adding temozolomide and radiotherapy in patients with newly-diagnosed glioblastoma.

The number of patients to be recruited is 30 over 6 months at 8 sites specialising in neuro-oncology.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and sign the informed consent document
* Men or women ≥18 years and ≤70 years
* Newly-diagnosed GB confirmed by biopsy or by resection in the 4-7 weeks before being registered in the trial.
* Patients must have at least 15 slides without staining or a tissue block (frozen or paraffin-embedded) available from a previous biopsy or surgery (tumour sample previously archived).
* Patients must have recovered from previous surgeries (time between surgery and inclusion in the study: 6 weeks).
* Karnofsky Index ≥60%.
* Adequate bone marrow reserve: haemoglobin ≥10 g/dL, WBC >3,000/mcL, absolute neutrophil count (ANC) ≥1,500 cells/μL, platelets ≥100,000 cells/μL.
* Adequate liver function: Bilirubin <1.5 times the upper limit of normal (ULN); AST ≤2.5 x ULN
* Creatinine clearance >60 ml/min/1.73 m2.
* The study treatment's effects on the development of the human foetus are not known. For this reason, women of childbearing age and men must agree to use a suitable birth control method (hormonal, barrier, abstinence or surgical sterilisation) before inclusion in the study, for the duration of the study and for at least 3 months after completing the trial treatment. The definition of an effective method of birth control is based on the judgement of the principal investigator or their designee. If a woman is pregnant or there is suspicion that she might be pregnant while participating in the study, she must inform the trial doctor immediately. All women of childbearing age should have a negative pregnancy test (serum/urine) in the 2 weeks prior to the beginning of treatment.

Exclusion Criteria:

* Presence of extracranial metastatic disease.
* Any previous treatment for glioblastoma.
* Patients who have had a Gliadel implant in the surgery.
* Use of an enzyme-inducing antiepileptic drug. Patients receiving this type of drug must have a washout period of at least 7 days prior to study inclusion.
* Previous abuse of cannabinoids.
* Presence of any clinically significant gastrointestinal abnormality that may affect the intake, transit or absorption of the study drug, such as the inability to take medication in the form of oral tablets or solution.
* Presence of any psychiatric or cognitive impairment that limits understanding or the signing of the informed consent and/or compromises compliance with the requirements of this protocol.
* Significant or uncontrolled cardiovascular disease, including: 1. Myocardial infarction in the previous 12 months. 2. Uncontrolled angina in the previous 6 months. 3. Congestive heart failure in the previous 6 months. 4. Diagnosed or suspected congenital long QT syndrome. 5. History of ventricular arrhythmias of any clinically significant type (such as ventricular tachycardia, ventricular fibrillation or torsades de pointes). 6. QTc prolongation on an electrocardiogram prior to entry (>470 ms). 7. History of second- or third-degree heart block (these patients may be eligible if they carry pacemakers). 8. Heart rate <50/min on the baseline electrocardiogram. 9. Uncontrolled hypertension
* Any patient with a history of significant cardiovascular disease, even if it is currently controlled, or who presents signs or symptoms that suggest impaired left ventricular function according to the investigator should have an assessment of left ventricular ejection fraction (LVEF) by ECCO or MUGA. If the LVEF in these circumstances is below the site's lower limit of normality or less than 50%, the patient will not be eligible.
* History of any cancer, except in the following circumstances: Patients with a history of other malignancies are eligible if they have been disease-free for at least the last 3 years and if, in the investigator's opinion, there is a low risk of disease recurrence. People with the following cancers are eligible, even if they have been diagnosed and treated in the past 3 years: cervical carcinoma in situ and basal cell carcinoma.

Patients will not be eligible if there is evidence of another cancer that required therapy other than surgery in the past 3 years.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-08-18 (Actual); Primary Completion 2025-11-13 (Actual); Study Completion 2025-11-13 (Actual)

PRIMARY OUTCOMES:
THC-CBD Maximum tolerated dose | 9 weeks
  After intra-patient dose escalation period, recommended dose of Glasdegib administeres with temozolamide during and after RT.
Incidence of Treatment-Emergent Adverse Events | 12 months
  Type and number or adverse events reported during THC-CBD treatment, based on the CTCAE reference criteria.

SECONDARY OUTCOMES:
Antitumor activity of THC-CBD combination with temozolamide and radiotherapy | 12 months
  Based on the tumor response in patients with measurable disease, after comparison of baseline characteristics and follow-up evaluations
Overall survival | 12 months
  Time between the start of treatment to death
Progression free survival | 12 months
  Time between the start of treatment and progression of disease
Expression of Midkine | 12 months
  Correlation of expression of midkine in peripheral blood and response to the experimental treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Benavides, M.D., Ph.D., Principal Investigator — Hospital Universitario y Regional de Málaga y Virgen de la Victoria
Locations (8):
- Spain (8):
  - Hospital Universitario Virgen del Rocío, Seville, Andalusia
  - Institut Català d'Oncología L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Son Espases, Palma de Mallorca, Mallorca
  - Hospital del Mar, Barcelona
  - Complejo Hospitalario Regional Virgen de las Nieves, Granada
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Clínico Universitario de Salamanca, Salamanca

IPD SHARING:
Plan to Share IPD: Undecided